CLINICAL TRIAL: NCT01310634
Title: Epidemiology and Prevention of Anxiety and Depression in Parents of Hospitalized Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Director, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMU-FY2011-236
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: Neonates; Parenting; Anxiety; Depression
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive intervention (Experimental): Parents of hospitalized neonates received Comprehensive intervention program.
  Interventions: Behavioral: Comprehensive intervention
- Conventional treatment (Other): Usual educational program
  Interventions: Behavioral: Comprehensive intervention

INTERVENTIONS:
Behavioral: Comprehensive intervention — Parents of hospitalized neonates received comprehensive intervention program,including parent educational-behavioral intervention program, effective doctor/nurse parent communication,regularly visit the neonatal ward and care the hospitalized neonates under the guidance of a doctor.
  Other Names: Comprehensive intervention program.

SUMMARY:
The overall goal of this project is to elucidate the epidemiology of anxiety and depression in parents of hospitalized neonates and test a comprehensive intervention program to prevent anxiety and depression in parents in this setting.

DETAILED DESCRIPTION:
Parents of hospitalized neonates experience high stress levels and feelings of helplessness in the neonatal ward and often concern for the health and well being of their fragile infant. Parental stress associated with admission to the neonatal ward of infants has been extensively studied in developed countries for many years, but rarely have epidemiological and intervention studies been reported in Chinese parents of hospitalized neonates. The aim of the present study was to elucidate the epidemiology of anxiety and depression in parents of hospitalized neonates and test a comprehensive intervention program to prevent anxiety and depression in parents in a Chinese hospital.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and reads Chinese
* No severe handicapping conditions or mental diseases
* Informed consent, no medical dispute
* Infants born within 28 days to be cared in the neonatal ward for at least 24 hours

Exclusion Criteria:

* Significant mental health history
* Newborns died within a week after hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Parental anxiety symptoms | 3 weeks
  Parents of Hospitalized Neonates were asked to complete the Self-rating Anxiety Scale (SAS) at 3 weeks after enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Shuping Han, PhD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Kong LP, Cui Y, Qiu YF, Han SP, Yu ZB, Guo XR. Anxiety and depression in parents of sick neonates: a hospital-based study. J Clin Nurs. 2013 Apr;22(7-8):1163-72. doi: 10.1111/jocn.12090. PMID 23480505